CLINICAL TRIAL: NCT05152069
Title: Spatio-temporal Parameters of Walking in Patients Hospitalized in Acute Geriatrics: Comparison of a Population of Fallers and Non-fallers
Brief Title: Spatio-temporal Parameters of Walking in Patients Hospitalized in Acute Geriatrics
Acronym: PST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8475
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Difficulty Walking
Keywords: Difficulty Walking; Elderly person; Spatio-temporal parameters
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of walking disorders in the elderly is high. These can lead to falls which represent a major public health issue in terms of hospitalization, morbidity and cost. Numerous studies analyzing the link between spatio-temporal parameters of gait and fall have already been carried out, but most have been carried out in a population of elderly patients living at home and having no or few comorbidities. Very few studies have been carried out in a population of frail elderly people, with multiple comorbidities or multiple medication, which is the case with most patients hospitalized in acute geriatrics.

The objective of the study is to evaluate the spatio-temporal parameters of walking using the GAITRite® mat in patients hospitalized in acute geriatrics and to compare them between a population of falling patients and a population of patients. no faller.

ELIGIBILITY:
Inclusion criteria:

* Subject aged > 70 years
* Have been hospitalized in an acute geriatric ward at the University Hospitals of Strasbourg between 01/06/2019 and 28/02/2020
* Have been able to walk on a square surface at least 12 meters long, with or without technical assistance
* Subject not having expressed, after being informed, his opposition to the reuse of his medical data for scientific research purposes.

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Non-autonomous subject for transfers and trips
* Subject under guardianship, curatorship or safeguard of justice

Min Age: 71 Years | Sex: All
Age Groups: Older Adult
Study Population: Subject aged > 70 years have been hospitalized in an acute geriatric ward at the University Hospitals of Strasbourg between 01/06/2019 and 28/02/2020 and ave been able to walk on a square surface at least 12 meters long, with or without technical assistance
Sampling Method: Non-Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05-24 (Estimated)

PRIMARY OUTCOMES:
Study of the spatio-temporal parameters of walking using the GAITRite® mat in patients hospitalized in acute geriatrics and to compare them between a population of falling patients and a population of patients. no faller. | Files analysed retrospectively from June 1, 2019 to February 28, 2020 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gériatrie Aigue - Hôpitaux Universitaires de Strasbourg, Strasbourg, France